CLINICAL TRIAL: NCT06082726
Title: The Systemic Availability of Short-Chain Fatty Acids After Delivery in the Small Intestine and the Colon
Brief Title: The Systemic Concentration of Short-Chain Fatty Acids After Delivery in the Small and Large Intestine of Healthy Volunteers
Acronym: Sistine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kristin Verbeke, Prof., KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: S67256
Record Dates: First submitted 2023-10-09; First posted 2023-10-13 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Systemic Availability; Intestinal Absorption; Metabolism; Short-chain Fatty Acids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- small intestinal delivery capsules (Experimental): Participants will ingest small intestinal delivery capsules filled with short-chain fatty acids.
  Interventions: Dietary Supplement: SCFA
- Colon-delivery capsules (Experimental): Participants will ingest colon-delivery capsules filled with short-chain fatty acids.
  Interventions: Dietary Supplement: SCFA

INTERVENTIONS:
Dietary Supplement: SCFA — Participants will ingest the capsules during a standard no fiber breakfast. A primed continuous infusion containing SCFA will run during the whole test day. Blood sampling will continue for 12 hours.

SUMMARY:
The goal of this crossover study is to evaluate the systemic availability of short-chain fatty acids (SCFA) that are either administered in the small intestine or the colon in healthy volunteers. The main question it aims to answer is whether the site of administration affects the amount of SCFA that reaches the systemic circulation. On two test days participants will ingest capsules filled with SCFA that are specifically delivered in the small intestine or the colon. After ingestion, blood samples will be collected at regular time points.

ELIGIBILITY:
Inclusion Criteria:

* female and male
* healthy participants
* age within 18 - 50 years
* normal BMI (18.5-25 kg/m^2)

Exclusion Criteria:

* Chronic gastrointestinal disorders such as inflammatory bowel disease (IBD), irritable bowel syndrome (IBS), celiac disease, chronic constipation (less than 3 stools a week) and chronic frequent diarrhoea (more than 3 stools a day)
* Previous abdominal surgery, except from appendectomy
* Being on a weight loss, gluten-free, lactose-free, or vegan diet
* The donation of blood during the last 3 months or suffering from low blood haemoglobin levels
* The use of antibiotics or other medication that affects the gastrointestinal tract 3 months preceding the study and/or during the study
* The use of prebiotics or probiotics 2 weeks preceding the study and/or during the study
* Pregnancy, lactation or wish to become pregnant during the study period
* Previous or current substance/alcohol dependence or abuse (> 2 units per day/14 units per week)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Estimated)
Dates: Start 2023-10-09 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Concentration of 13C-short-chain fatty acids in blood | up to 12 hours
  Assessed by analysing SCFA in blood samples collected at regular time points

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No
No IPD data will be shared with other researchers.